CLINICAL TRIAL: NCT05055596
Title: Improving Quality of Life for Adults Living With HIV and Chronic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23AT010099 (NIH); K23AT010099 (NIH)
Record Dates: First submitted 2021-09-02; First posted 2021-09-24 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections; Chronic Pain
MeSH Terms: conditions — HIV Infections; Chronic Pain | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentle Movement (Experimental)
  Interventions: Behavioral: Tai Chi
- Health Coaching (Active Comparator)
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Tai Chi — Qigong/Tai Chi Easy is a manualized intervention with formal training for instructors through the Institute of Integral Qigong and Tai Chi (IIQTC). The protocol can be modified based on participant needs and physical abilities. Qigong/Tai Chi Easy uses a series of repeated and simple-to-learn movements (rather than long forms with complicated choreography).
  Arms: Gentle Movement
Behavioral: Health Coaching — The Health Education group will be adapted from a previously developed time and attention control condition used in HIV research. Additional health education material will be based on information learned in the qualitative interviews conducted prior to the start of this study. Examples of session material include the following: sleep hygiene, healthy diet, sun safety, and healthy homes.
  Arms: Health Coaching

SUMMARY:
Chronic pain is highly comorbid among the 1.2 million persons living with HIV, with recent prevalence estimates ranging from 55-67%. Needed are evidenced-based non-pharmacological interventions to improve chronic pain management and reduce the demand for opioids in the United States. The proposed research will address this need by examining the feasibility and acceptability of Tai Chi as a mind-body intervention for chronic pain management in an HIV population.

DETAILED DESCRIPTION:
Persons living with HIV (PLWH) are at increased risk for chronic pain conditions, with prevalence rates estimated to be between 55-67%. While acute pain is a life-sustaining biological response to tissue damage or injury, chronic pain is a separate condition that often causes significant physical and psychological suffering. Causes of chronic pain among PLWH include disease progression, the impact of the virus on immune and nervous system function, and medication side-effects. PLWH, like many other chronic pain patients, may be prescribed opioid medications, which have not been found to be effective in managing non-cancer related chronic pain. Additionally, the significant risk of dependence and overdose far outweigh the potential benefit of opioid medications for chronic pain. Governing bodies in medicine have called for non-pharmacological interventions to be considered front-line treatment recommendations for chronic pain management. Mind-body interventions, such as mindfulness, yoga, and Tai Chi, have been shown to be effective at reducing pain symptoms and improving psychological outcomes for individuals with chronic pain. Unfortunately, few studies have examined the use of mind-body interventions for chronic pain management for PWLH, with even fewer using formative research to modify interventions to meet the unique needs of this vulnerable population. The research plan proposed in this application will address these gaps in the literature. This study will examine the feasibility and acceptability of a mind-body intervention, Qigong/Tai Chi Easy, for chronic pain management among PLWH. The researchers will recruit 40 individuals from the Comprehensive HIV Program at Temple Health. Following informed consent, participants will be randomized to mind-body arm or health education control arm. Participants in both arms will complete baseline assessment followed by a 10-week intervention. The mind-body intervention group will meet weekly for 60-minute sessions and be provided with a video for at-home practice. The health education group will also meet weekly for 60 minutes and be assigned weekly homework related to the topics discussed in session. At the conclusion of the 10 weeks, participants will complete at post-intervention assessment. A 3-month follow up assessment will also be completed. In addition to feasibility (i.e., recruitment rates, retention) and acceptability (i.e., satisfaction ratings), the researchers will assess pain symptoms (general and specific), perceived stress, depression, quality of life, and HIV medication adherence. The researchers anticipate that the study will demonstrate feasibility and acceptability as evidenced by adequate enrollment, retention, and satisfaction. Findings from the proposed study will be used to inform a future research grant with power to detect efficacy of the mind-body intervention for chronic pain management.

ELIGIBILITY:
Inclusion Criteria:

* age 45 and older;
* HIV positive status based on clinical records;
* chronic pain condition based on clinical records;
* English speaking;
* physically able to participate in a Tai Chi program

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Inability or unwillingness to travel to Temple Dental School;
* Inability or unwillingness to engage in 10-week intervention;
* Non-English speaking;
* Active substance use disorder;
* Acutely suicidal or psychotic;
* Self-reported participation in another research study related to chronic-pain

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain Rating (VAS) | Each intervention group session (10 weeks)
  Participants will be asked to rate their pain on a visual analog scale (ranging from 0, no pain, to 100, most extreme pain)
Brief Pain Inventory - Short Form (BPI) | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  A self-report of pain intensity, impairment in mobility, impairment in activities of daily living, mood, and pain-related anxiety/fear
Subjective Peripheral Neuropathy Screen Questionnaire (SPNSQ) | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  A valid and reliable measure of neuropathic pain symptoms for PLWH
Orebro Musculoskeletal Pain Screening Questionnaire (OMSPQ) | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  Measure used to assess musculoskeletal pain, with questions related pain site, and duration

SECONDARY OUTCOMES:
Quality of Life (WHO-QOL-BREF) | Baseline (Week 0), Post-Intervention (Weeks 10-12), and 3-month Follow Up (Weeks 22-24)
  Measure to assess feelings regarding quality of life, health, or other areas of one's life
Perceived Stress Scale (PSS) | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  Measure to assess frequency and severity of stressful situations, which may be relevant for people living with HIV and chronic pain as they manage intersecting chronic illnesses
Patient Health Questionnaire (PHQ-8) | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  The PHQ-9 is a commonly used measure of depression with strong psychometric properties for clinical populations
Pain Catastrophizing Scale (PCS) | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain.
The Meditative Movement Inventory | Post-Intervention (Weeks 10-12)
  This is a 17-item questionnaire aiming to capture in descriptions different aspects of meditative movement, such as the meditative state of mind, breathing, flow of movement and affective quality.
The HIV Medication Adherence Survey | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  Medication adherence will be assessed using a validated brief 3-item measure for PLWH, which assesses number of days missed, difficulty following instructions, and self-rating of medication adherence in the past 30 days

OTHER OUTCOMES:
Feasibility | Baseline (Week 0), Post-Intervention (Weeks 10-12), 3-month Follow Up (Weeks 22-24)
  Ability to recruit and retain participants through intervention and follow-up assessments
Acceptability | Post-Intervention (Weeks 10-12)
  Participant self-reported satisfaction with intervention components

CONTACTS AND LOCATIONS:
Overall Officials: Eugene M Dunne, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University Kornberg School of Dentistry (TUKSoD), Philadelphia, Pennsylvania, United States